CLINICAL TRIAL: NCT05925231
Title: Variability of Healthy People and People After Stroke Results in the Box and Block Test
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Rybářová, Occupational therapist, Charles University, Czech Republic
Other Study IDs: 75/23 S-IV
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Motor Activity
Keywords: Box and Block Test; Stroke; Czech Extended Version of Manual for the Box and Block Test
MeSH Terms: conditions — Motor Activity; Stroke | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People after stroke: Czech people after stroke, aged 20 - 64 years
  Interventions: Diagnostic Test: Box and Block Test
- Healthy population: Czech healthy people, aged 20 - 64 years
  Interventions: Diagnostic Test: Box and Block Test

INTERVENTIONS:
Diagnostic Test: Box and Block Test — 3 attempts of each subtest of the Box and Block Test performed according to the Czech Extended Version of Manual for the Box and Block Test
  Other Names: questionnaire

SUMMARY:
Main aim of the study is to find out how many attempts of each subtest in the Box and Block Test should be done in clinical practice during testing people after stroke who are 20-64 years old.

ELIGIBILITY:
Inclusion Criteria:

* people after stroke 20 - 64 years old
* signed Informed consent for probation with inclusion to research and Consent to the collection and processing of personal data during the study at the General University Hospital in Prague
* ability to sit independently for 15 minutes
* ability to grasp and move at least one 25 mm wide cube placed on a table using the dominant and then the non-dominant upper limb across the test partition
* ability to perform a simple task following verbal instructions
* retained ability to understand - according to psychological examination
* completion of testing during hospitalization in the Beroun Rehabilitation Hospital

Exclusion Criteria:

* severe hearing impairment not corrected by a hearing aid
* severe visual impairment not corrected by glasses
* severe comprehension impairment
* other reasons not allowing the completion of the entire testing using the Box and Block Test

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People after stroke, healthy people
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
results from the Box and Block Test | 30 minutes
  number of transported blocks

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Rehabilitation Hospital of Beroun, Beroun
  - Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: No